CLINICAL TRIAL: NCT01418859
Title: Status and the Application of Topotecan at Post-operation Treatment of Cervical Cancer
Brief Title: Clinical Study in Post-operation Treatment of Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Liu Zi, Profesor, Xi'an Jiaotong University
Other Study IDs: GCR-01
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; postoperation; chemotherapy; radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- radiation therapy only: Including criteria: cervical cancer patients after surgery with big tumor, deep invasion or tumor thrombi in the vascular system, but without lymph invasion, positive surgery margin or parametrium invasion. Patients in this group receive radiation therapy only. radiation therapy regimen: 3D-CRT pelvic radiation, 95%CTV DT 45Gy/25f. Radiation field include tumor bed and regional lymph nodes area. Upper border: branching of abdominal aorta. The radiation fields go down along the iliac vessels (including regions of 7mm out of the iliac vessels) and include the tumor bed region. Lower border: the inferior margin of obturator foramen.
- concurrent chemoradiotherapy: Including criteria: cervical cancer patients after surgery with big tumor, deep invasion or tumor thrombi in the vascular system, but without lymph invasion, positive surgery margin or parametrium invasion. Patients in this group receive concurrent chemotherapy and radiation therapy. radiation therapy regimen is the same with radiation therapy only group. Chemotherapy regimen: Topotecan (1.5mg /m2 d1,2, 1mg d3) and Cisplatin (25mg /m2 d1-3). Chemotherapy will be carry out in the 2nd and 6th week of radiation therapy.
- concurrent and additional chemotherapy: Including criteria: cervical cancer patients after surgery with big tumor, deep invasion or tumor thrombi in the vascular system, but without lymph invasion, positive surgery margin or parametrium invasion. Patients in this group receive concurrent chemotherapy and radiation therapy, and additional chemotherapy after concurrent treatment. radiation therapy regimen is the same with radiation therapy group. Chemotherapy regimen: Topotecan (1.5mg /m2 d1,2, 1mg d3) and Cisplatin (25mg /m2 d1-3). Chemotherapy will be carry out in the 2nd and 6th week of radiation therapy. Additional chemotherapy regimen is the same with concurrent chemotherapy, and will be carry out in the 4th and 8th week after radiation therapy.

SUMMARY:
The purpose of the research is to evaluate the effect of additional chemotherapy in postoperation therapy of cervical cancer patients with risk factors (big tumor, deep invasion or tumor thrombi in the vascular system).

DETAILED DESCRIPTION:
Cervical cancer has a very high morbidity. Many patients need additional therapy after surgery in order to elevate the survival rate and life quality. In this research, we are going to give additional therapy to patients who have big tumor, deep invasion or tumor thrombi in the vascular system after surgery. randomized control method will be used in this research, in order to compare the survival rate and side effects between radiation therapy only, concurrent chemoradiotherapy, and concurrent chemoradiotherapy with additional chemotherapy. 3D-CRT and Topotecan will be used in this research.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent the cervical cancer radical surgery in three months have higt risk factors which including deep stromal invasion,large primary tumour and/or lymphovascular spase invasion;
2. squamous carcinoma;
3. age<70;
4. Gynecologic Oncology Group (GOG):0-2.

Exclusion Criteria:

1. negative nodes,surgical margin,and/or parametrium;
2. No serious damage to the liver and kidney function, no hypertension,diabetes and other effects of therapy complications.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent the cervical cancer radical surgery in three months have higt risk factors which including deep stromal invasion,large primary tumour and/or lymphovascular spase invasion.
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chen M W, M.D, Study Director — Affiliated Hospital of Medical College of Xo'an Jiaotong University
Locations (1):
- Xi'an Jiaotong University College of Medicine, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Sun W, Wang T, Shi F, Wang J, Wang J, Hui B, Zhang Y, Lu J, Chen H, Liu Z. Randomized phase III trial of radiotherapy or chemoradiotherapy with topotecan and cisplatin in intermediate-risk cervical cancer patients after radical hysterectomy. BMC Cancer. 2015 May 4;15:353. doi: 10.1186/s12885-015-1355-1. PMID 25935645